CLINICAL TRIAL: NCT02236390
Title: Integrating Sleep and PTSD Treatment: Examining the Role of Emotion Regulation
Brief Title: Integrating Sleep, Nightmare and PTSD Treatments
Acronym: CPTERRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Joanne Davis, Professor, University of Tulsa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU1459R1; HR14-127 (Other Grant/Funding Number: OCAST)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Nightmares; PTSD
Keywords: Nightmare; PTSD; Sleep; Emotion Regulation; Exposure Relaxation and Rescripting Therapy; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Processing Therapy-Cognitive (Active Comparator): 12 sessions of cognitive processing therapy-Cognitive
  Interventions: Behavioral: Cognitive Processing Therapy - Cognitive
- ERRT + CPT-C (Active Comparator): 5 sessions of Exposure, Relaxation, and Rescripting Therapy, followed by 12 sessions of Cognitive Processing Therapy- Cognitive
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy; Behavioral: Cognitive Processing Therapy - Cognitive
- CPT-C + ERRT (Active Comparator): 12 sessions of Cognitive Processing Therapy - Cognitive, followed by 5 sessions of Exposure, Relaxation, and Rescripting Therapy
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy; Behavioral: Cognitive Processing Therapy - Cognitive

INTERVENTIONS:
Behavioral: Exposure, Relaxation, and Rescripting Therapy — 5 sessions that last approximately one hour addressing nightmares and sleep problems. Participants will log sleep events and associated symptoms
  Other Names: ERRT; IRT
  Arms: CPT-C + ERRT; ERRT + CPT-C
Behavioral: Cognitive Processing Therapy - Cognitive — 12 sessions cognitive behavioral treatment targeting posttraumatic stress symptoms.
  Other Names: CPT-C; CPT

SUMMARY:
The purpose of the proposed pilot study is to extend previous findings regarding the efficacy of a brief treatment for chronic posttrauma nightmares and sleep problems by integrating this treatment with evidence-based treatment for posttraumatic stress disorder (PTSD). Cognitive processing therapy (CPT) (Resick & Schnicke, 1996) is a well-established and efficacious evidence-based psychological treatment for PTSD in both civilian and veteran populations (Forbes et al., 2012; Monson et al., 2006; Resick et al., 2008; Resick, Nishith, Weaver, Astin, & Feuer, 2002). The U.S. Department of Veterans Affairs (VA) includes CPT among the first-line treatments for PTSD (National Center for PTSD, 2012). A modified protocol without the utilization of written exposure (CPT-C) may be more effective than the original protocol. However, despite such promising evidence, individuals who experience chronic nightmares and sleep problems tend to show smaller gains and persistent nightmares following PTSD treatment (Nappi, Drummond, & Hall, 2012). Given that nightmares are considered the hallmark of PTSD (Ross, Ball, Sullivan, & Caroff, 1989) and their treatment-resistant nature (Davis & Wright, 2007), specific psychological treatments have been developed to target sleep disturbances and nightmares.

Exposure, relaxation, and rescripting therapy (ERRT) is a promising psychological intervention developed to target trauma-related nightmares and sleep disturbances. Though further evidence is needed, ERRT has exhibited strong support in reducing the frequency and intensity of nightmares, as well as improving overall sleep quality in both civilian and veteran samples. In addition, significant decreases in PTSD and depression symptoms have been reported following treatment (Davis et al., 2011; Davis & Wright, 2007; Long et al., 2011; Swanson, Favorite, Horin, & Arnedt, 2009). ERRT is currently an evidence-level B suggested treatment (Cranston, Davis, Rhudy, & Favorite, 2011).

There is a call to research suggesting the importance of treatment studies which focus on interventions that integrate nightmare and sleep symptom treatment with evidence-based treatment for PTSD (Nappi et al., 2012). In an effort to respond to this call, we propose to tailor ERRT for use in conjunction with CPT, and preliminarily test ERRT's additive effect to CPT in treating PTSD in community outpatients. We hypothesize that ERRT would increase CPT's treatment efficacy by its specific focus on trauma-related nightmares and sleep disturbances. Sleep difficulties are known to increase tension, and reduce one's ability to cope adaptively (Bonn-Miller, Babson, Vujanovic, & Feldner, 2010; Hofstetter, Lysaker, & Mayeda, 2005; Nishith, Resick, & Mueser, 2001). Thus, with improved sleep an individual may have additional personal coping resources for which s/he can use to address the broader trauma issues (Nappi et al., 2012). To test this integration, we will compare ERRT + CPT, CPT + ERRT, and CPT alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of Age minimal
* Experienced a trauma
* One nightmare per week for past month, minimal
* meet full criteria for PTSD

Exclusion Criteria:

* 17 years of age or younger
* acute psychosis
* bipolar disorder
* intellectual disability
* active suicidality
* untreated substance use disorder within past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-08; Primary Completion 2024-11 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Nightmare Frequency | up to 6-months follow-up
  A fill-in-the blank question (range = 0-X nightmares) from the Trauma Related Nightmare Survey will be utilized to determine the past week nightmare frequency at baseline, and 3 and 6 months follow-up. Higher values indicate more nightmares.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale | Past Month symptoms measured at baseline, and 3 and 6 month follow-up
  This semi-structured clinical interview assesses severity of each of 30 items measuring Diagnostic and Statistical Manual (DSM-5) criteria for PTSD on a 5-point scale (0 - 4), (possible range: 0-80). A symptom is considered present if the severity is rated 2 or higher. Total scores are comprised of four factors (reexperiencing, avoidance, cognitive/emotional and hyperarousal)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne l Davis, PhD, Principal Investigator — University of Tulsa
Locations (1):
- University of Tulsa, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Davis JL, Rhudy JL, Pruiksma KE, Byrd P, Williams AE, McCabe KM, Bartley EJ. Physiological predictors of response to exposure, relaxation, and rescripting therapy for chronic nightmares in a randomized clinical trial. J Clin Sleep Med. 2011 Dec 15;7(6):622-31. doi: 10.5664/jcsm.1466. PMID 22171201
- See also: Related Info — http://nightmaretreatment.org